CLINICAL TRIAL: NCT05415371
Title: Monetary Incentives to Promote Engagement With the Oklahoma Tobacco Helpline Among Pregnant Women With Medicaid
Brief Title: Persistent Poverty Counties Pregnant Women With Medicaid
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14736
Record Dates: First submitted 2022-05-25; First posted 2022-06-13 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Tobacco Cessation; Tobacco Use; Tobacco Smoking; Smoking Cessation Financial Incentives; Socioeconomic Status; Contingency Management; Pregnancy
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use; Tobacco Smoking | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Participants randomized to Standard Care will be offered weekly counseling calls and pharmacotherapy.
  Interventions: Other: Standard Care
- Standard Care + Financial Incentives (Experimental): Financial Incentives participants will receive standard care plus incentives for completing counseling calls and abstinence.
  Interventions: Behavioral: Standard Care + Financial Incentives; Other: Standard Care

INTERVENTIONS:
Behavioral: Standard Care + Financial Incentives — Financial incentive participants will receive standard care and receive incentives for completing counseling calls and for abstinence.
  Arms: Standard Care + Financial Incentives
Other: Standard Care — Participants randomized to Standard Care will be offered weekly counseling calls and pharmacotherapy.

SUMMARY:
Although many women initially quit smoking during pregnancy, most will return to smoking by the end of pregnancy or during the first 6 months postpartum. The proposed pilot project is designed to evaluate the feasibility and potential efficacy of offering small financial incentives for the completion of smoking cessation coaching and biochemically-verified smoking abstinence at follow-up among pregnant women with Medicaid insurance who contact the Oklahoma Tobacco Helpline (OTH). The study will enroll 100 pregnant women who will be randomly assigned to OTH care or OTH plus escalating incentives (OTH+I) for completing up to 5 coaching calls over the first 8 weeks after enrolling (prepartum) and for biochemically-verified smoking abstinence at 9 weeks post-enrollment (assessed remotely via smartphone). In addition, participants will be incentivized for completing a postpartum coaching call by 8 weeks postpartum. Feasibility outcomes for the incentives based intervention will focus on coaching call completion, rates of prepartum and postpartum follow-up, biochemically-verified smoking cessation, and perceptions of the intervention. Potential effectiveness will be evaluated by comparing biochemically-verified smoking abstinence rates in OTH+I relative to OTH alone at 12 weeks post-enrollment (prepartum) and 12 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria

* contact the Oklahoma Tobacco Helpline seeking smoking cessation treatment, and enroll in the multiple call program
* are a female ≤ 25 weeks pregnant
* report smoking ≥ 5 cigarettes per day
* are ≥ 18 years of age
* are able to provide a copy/photo of their ID/driver's license or other documentation of identity
* are able to read, speak, and understand English

Exclusion Criteria

• participants will be excluded if they do not meet the inclusion criteria

Ages: 18 Years to 105 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically verified abstinence 12 weeks post enrollment | 12 weeks post enrollment
  The outcome measure is biochemically verified over 7-day point prevalence at 12 weeks post-enrollment.
Self-reported abstinence 12 weeks postpartum | 12 weeks postpartum
  The outcome measure is biochemically verified abstinence over 7-day point prevalence at 12 weeks post-partum

CONTACTS AND LOCATIONS:
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States